CLINICAL TRIAL: NCT02729233
Title: Predicting Clinical Response to Golimumab With Mucosal Barrier Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: University of Arkansas (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 205241
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Ulcerative Colitis
Keywords: mucosal barrier function
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients receiving biopsies (Other): UC patients who will be started on golimumab for treatment of UC (moderate to severe flare, steroid dependence, or failure of other therapies), epithelial barrier function will be characterized using probe-based confocal laser endomicroscopy (pCLE).
  Interventions: Other: patients receiving biopsies

INTERVENTIONS:
Other: patients receiving biopsies — Six mucosal biopsies will be collected from each site (terminal ileum and rectum) for histologic verification of pCLE findings at baseline, and again at month 12 for a total of 12 research samples per colonoscopy, or 24 research biopsy samples during the course of the study. The study subjects will be followed for a total of 1 year after initial colonoscopy with pCLE. The primary study end-point is clinical response at 3 months following initiation of golimumab.

SUMMARY:
Ulcerative colitis (UC) is a chronic relapsing inflammatory bowel disease (IBD). UC is an ongoing disease of the colon or large intestine. Studies have shown that leakiness of the gut plays a major role in the development of UC. Leakiness of the gut is a condition that is a result of damage to the intestinal lining, making it less able to protect its internal environment as well as to filter needed nutrients and other substances. Some bacteria, toxins, and waste not normally absorbed may get into the blood stream.

Golimumab is an FDA approved medication used for the treatment of moderate to severe ulcerative colitis. The investigators have evidence to suggest that measuring the leakiness of the gut using a tool called a confocal laser endomicroscope may be able to predict how well a patient's body will respond to treatment of UC with golimumab. Confocal laser endomicroscopy (CLE) is an FDA approved technique that can look at the cells of a patient's gut during colonoscopy to assess the leakiness of gut.

The objective of this study is to determine how the leakiness of the gut in patients with UC can predict response to golimumab therapy.

DETAILED DESCRIPTION:
The objective of this pilot study is to determine the predictive value of mucosal barrier dysfunction for a therapeutic response to golimumab in UC patients. This objective is based on the investigator's hypothesis that barrier dysfunction is a potent predictor of response to anti-tumor necrosis factor (TNF) therapy. This hypothesis is based on the following observations: (1) IBD patients with higher gap densities have higher mucosal pro-inflammatory cytokine levels; (2) the highest rates of response to biologic therapy for Ulcerative colitis are seen in post-operative patients, with over 90% endoscopic remission rate at one year; and (3) prominent barrier dysfunction is observed at the anastomotic site in animal models of ileal resection. Therefore, the investigators hypothesize that barrier dysfunction is a potent predictor of therapeutic response to golimumab in UC patients.

In 30 UC patients who will be started on golimumab for treatment of UC (moderate to severe flare, steroid dependence, or failure of other therapies), epithelial barrier function will be characterized using probe-based CLE (pCLE). Six mucosal biopsies will be collected from each site (terminal ileum and rectum) for histologic verification of pCLE findings at baseline, and again at month 12 for a total of 12 research samples per colonoscopy, or 24 research biopsy samples during the course of the study. The study subjects will be followed for a total of 1 year after initial colonoscopy with pCLE. The primary study end-point is clinical response at 3 months following initiation of golimumab.

Secondary study endpoints are: (1) The rate of clinical remission at 3 months following initiation of golimumab. (2) The rate of clinical remission at 12 months following initiation of golimumab. (3) Endoscopic and histological evidence of mucosal healing at one-year follow-up colonoscopy.

Clinical Response & Remission definitions are: (1) Clinical Remission: partial Mayo score of 2 points, without any sub-score >1. (2) Clinical Response: reduction of partial Mayo UC score by ≥ 30% and ≥ 2 points, with a rectal bleeding sub-score of ≤ 1 or a decrease in the bleeding sub-score of ≥ 1.

Endoscopic and histologic mucosal healing definitions: (1) Endoscopic: Mayo endoscopic score of 0 or 1. (2) Histologic: Riley's histological score ≤ 6.

The investigators proposal is based on clinical, translational and basic evidence of barrier dysfunction in the pathogenesis of UC. With the development of a robust prediction model for therapeutic response, UC patients can be treated more effectively with golimumab. Using a stratified approach, higher therapeutic response rate may eventually yield a new "intelligent step-up" treatment strategy in this personalized medicine era.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ulcerative colitis based on standard clinical, radiological, endoscopic and histological criteria with moderate-to-severe disease activity, defined as a Mayo score of 6-12, with an endoscopic subscore of 2 or more.
2. Age 18-75 years
3. Patients about to be started on golimumab therapy because of moderate to severe flare, steroid dependence, or failure of other therapies.
4. Inadequate response to or failure to tolerate 1 or more of the following conventional therapies:

   * Oral 5-aminosalicylates (5-ASAs)
   * Oral corticosteroids
   * Immunosuppressives (azathioprine (AZA) or 6-mercaptopurine) OR
   * Corticosteroid-dependent (i. e., could not taper corticosteroids without recurrence of UC symptoms) AND
   * No previous exposure to biological therapy (TNF naïve)
5. Patients concurrently treated with oral 5-aminosalicylates or corticosteroids must have maintained stable dose for ≥ 2 weeks before baseline.
6. Patients concurrently treated with AZA and/or 6-mercaptopurine must have maintained stable dose for ≥ 4 weeks before baseline.
7. Tuberculosis (TB) related screening criteria:

   1. No history of latent or active tuberculosis (TB) prior to screening. An exception is made for subjects who have a history of latent TB and are currently receiving treatment for latent TB, will initiate treatment for latent TB prior to first administration of golimumab, or have documentation of having completed appropriate treatment for latent TB within 3 years prior to the first administration of golimumab.
   2. No signs or symptoms suggestive of active TB upon medical history and/or physical examination.
   3. No recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to the first administration of study agent.
   4. Within 2 months prior to the first administration of golimumab, have a negative QuantiFERON®-TB Gold test result, or have a newly identified positive QuantiFERON®-TB Gold test result in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated prior to the first administration of study agent. Subjects with persistently indeterminate QuantiFERON®-TB Gold test results may be enrolled without treatment for latent TB, if active TB is ruled out, their chest radiograph shows no abnormality suggestive of TB (active or old, inactive TB), and the subject has no additional risk factors for TB as determined by the principal investigator.
   5. Have a chest radiograph posterior-anterior views, taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current, active TB or old, inactive TB.

Exclusion Criteria:

1. Pregnancy/nursing.
2. Known allergies to IV contrast or shellfish.
3. Impaired renal function (serum creatinine over 1.5 mg/dL).
4. Uncontrolled or severe asthma.
5. Active infection.
6. Active or previously identified latent tuberculosis.
7. History of systemic lupus.
8. Current or history of demyelinating neurological disease.
9. Current or history of congestive heart failure.
10. History of or at imminent risk for colectomy.
11. Gastrointestinal surgery ≤ 2 months prior to screening for study entry.
12. Colitis limited to 20 cm. of the colon.
13. History of colonic mucosal dysplasia or adenomatous colonic polyps that were not removed.
14. Screening stool sample positive for enteric pathogens or Clostridium difficile toxin.
15. Previous use of the following medications:

    * Biologic anti-TNF agent(s) natalizumab or other agents targeting the α-4integrin, B-cell-depleting agents (rituximab) or T-cell-depleting agents (vedolizumab, visilizumab) within 12 months of study entry.
    * Continued B- or T-cell depletion ˃ 12 months after completing therapy with lymphocyte-depleting agents.
    * Oral corticosteroids at a dose ˃ 40 mg. prednisone or its equivalent per day
    * Use of cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 8 weeks of study entry.
    * Use of an investigational agent within 5 half-lives of that agent prior to study entry.
16. History of any malignancy.
17. History of active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening.
18. Subjects must undergo screening for hepatitis B virus (HBV). At a minimum, this includes testing for HBsAg (HBV surface antigen), anti-HBs (HBV surface antibody), and anti-HBc total (HBV core antibody total):

    1. Subjects who test negative for all HBV screening tests (ie, HBsAg-, anti-HBc-, and anti HBs-) are eligible for this study.
    2. Subjects who test positive for surface antigen (HBsAg+) are not eligible for this study, regardless of the results of other hepatitis B tests.
    3. Subjects who test negative for surface antigen (HBsAg-) and test positive for core antibody (anti-HBc+) and surface antibody (anti-HBs+) are eligible for this study.
    4. Subjects who test positive only for surface antibody (anti-HBs+) are eligible for this study.
    5. Subjects who test positive only for core antibody (anti-HBc+) must undergo further testing for hepatitis B deoxyribonucleic acid (HBV DNA test). If the HBV DNA test is positive, the subject is not eligible for this study. If the HBV DNA test is negative, the subject is eligible for this study. In the event the HBV DNA test cannot be performed, the subject is not eligible for this study.

1. Subjects with a positive HBV DNA test will be counselled per the clinical Hepatitis B Positive Screen Standard Operating Procedure (SOP). If the HBV DNA test cannot be performed, the subject will be counselled per the SOP at the physician's discretion.

19. Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening.

20. Have a chest radiograph within 3 months prior to the first administration of golimumab that shows an abnormality suggestive of a malignancy or current active infection, including TB.

21. Have had a nontuberculous mycobacterial infection or opportunistic infection (e. g., cytomegalovirus, pneumocystosis, aspergillosis) within 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Rate of improvement in mucosal barrier function as measured by pCLE | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia J Liu, MD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No